CLINICAL TRIAL: NCT03697304
Title: An Open-label, Phase II, Platform Trial Evaluating Safety and Efficacy of Multiple BI 754091 (Ezabenlimab) Anti-PD-1 Based Combination Regimens in PD-(L)1 naïve and PD-(L)1 Pretreated Patient Populations With Advanced and/or Metastatic Solid Tumours Who Have Had at Least One Line of Systemic Therapy
Brief Title: Platform Trial Evaluating Safety and Efficacy of Ezabenlimab Anti- PD-1 Based Combination Therapies in PD-(L)1 naïve and PD- (L)1 Pretreated Patient Populations With Advanced/Metastatic Solid Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1381-0009; 2018-002344-81 (EudraCT Number)
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Neoplasm Metastasis; Advanced Tumors; Metastatic Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Module C, Cohort 1: GEC patients (Experimental): Patients with locally advanced, unresectable or metastatic gastric adenocarcinoma or gastro-oesophageal adenocarcinoma (GEC) with at least one prior systemic treatment, who failed standard therapy, for whom no further effective options existed, and with no prior PD-1 or PD-L1-based treatment, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 720 mg of BI 836880, in the form of i.v. infusion, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 836880
- Module C, Cohort 2: 2ary resistance patients (Experimental): Patients with any advanced or metastatic solid tumor (excluding non-squamous lung cancer, non-small-cell lung cancer, and melanoma) who had received prior anti-PD-1- or anti-PD-L1-based treatment and progressed after achieving benefit (at least stable disease with a minimum duration of benefit of 4 months) and minimum treatment duration of 2 months on the previous anti-PD-1- or anti-PD-L1-based treatment without progressive disease, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 720 mg of BI 836880 on Day 1, intravenously, on Day1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 836880
- Module C, Cohort 3: 1ary resistance patients (Experimental): Patients with select advanced or metastatic solid tumors with prior anti-PD-1- or anti-PD-L1-based treatment without achieving benefit ( stable disease duration of less than 4 months or progressive disease in less than 4 months while on treatment), were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 836880
- Module C, Cohort 4: CRC patients (Experimental): Patients with locally advanced, unresectable or metastatic second-line or greater, microsatellite-stable colorectal cancer (CRC) without prior anti-PD-1- or anti-PD-L1-based treatment, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 836880
- Module C, Cohort 5: EC patients (Experimental): Patients with advanced endometrial carcinoma (EC), excluding microsatellite instability-high or mismatch repair deficient types, who progressed following one line of chemotherapy, were not eligible for curative surgery or radiation, and had not been previously treated with anti-PD-1- or anti-PD-L1-based therapies, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 836880
- Module A, Cohort 1: GEC patients (Experimental): Patients with locally advanced, unresectable or metastatic gastric adenocarcinoma or gastro-oesophageal adenocarcinoma, who received prior anti-PD-1 or anti-PD-L1-based treatment, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Module A, Cohort 2: 2ary resistance patients (Experimental): Patients with any advanced or metastatic solid tumors who had been previously treated with anti-PD-1 or anti-PD-L1-based therapies, and who progressed after achieving benefit (at least stable disease with a minimum duration of benefit of 6 months) and minimum treatment duration of 2 months without experiencing disease progression, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Module A, Cohort 3: 1ary resistance patients (Experimental): Patients with select advanced or metastatic solid tumor types, who have been previously treated with previous anti-PD-1 or anti-PD-L1-based therapies without achieving benefit (stable disease for less than 6 months or progressive disease in less than 6 months), were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along with 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111

INTERVENTIONS:
Drug: Ezabenlimab — 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles.
  Other Names: BI 754091
Drug: BI 754111 — 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
  Arms: Module A, Cohort 1: GEC patients; Module A, Cohort 2: 2ary resistance patients; Module A, Cohort 3: 1ary resistance patients
Drug: BI 836880 — 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
  Arms: Module C, Cohort 1: GEC patients; Module C, Cohort 2: 2ary resistance patients; Module C, Cohort 3: 1ary resistance patients; Module C, Cohort 4: CRC patients; Module C, Cohort 5: EC patients

SUMMARY:
This is a study in adults with various types of advanced cancer. The purpose of the study is to test a medicine called BI 754091 in combination with several other cancer medicines. BI 754091 is an immunotherapy. This means it may help the immune system fight cancer. Such therapies are also called immune checkpoint inhibitors.

How long the participants are in the study depends on whether they benefit from treatment and whether they experience unacceptable side effects. The participants are put into different groups. Each group receives BI 754091 in combination with another medicine.

The doctors check whether the tumors shrink or disappear. The doctors also check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria

Master Protocol:

* Provision of signed and dated, written Master informed consent form (ICF) prior to any trial-specific procedures, sampling, or analyses.
* Patient ≥18 years of age at the time of signature of the ICF.
* Eastern Cooperative Oncology Group (ECOG) score: 0 or 1.
* Patient must agree to a pre-treatment biopsy (if archival tissue is not available) and on-treatment tumour biopsy. If archived tumour tissue is available from the last treatment failure, sections may be supplied instead of a pre-treatment biopsy.
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be willing and able to use highly effective methods of birth control (that result in a low failure rate of less than 1% per year when used consistently and correctly) during trial participation and for at least 6 months after the last administration of trial medication. Acceptable highly effective methods of contraception include total sexual abstinence when this is in line with the preferred and usual lifestyle of the study participant (periodic abstinence such as calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception), an intrauterine device or intrauterine hormone-releasing system, bilateral tubal ligation, and vasectomised partner (with post-vasectomy proof of absence of sperm). Male patients with partners of childbearing potential must agree to use condoms and ensure their partners are using an additional highly effective method of birth control, during the trial and until at least 6 months after the end of the trial treatment.

Module A:

- Histologically confirmed diagnosis of one of the following cohorts:

* Cohort 1 GEC - Locally advanced, unresectable or metastatic gastric adenocarcinoma or gastro oesophageal adenocarcinoma (GEC) (defined as primary tumour localisation below the gastro oesophageal junction (GEJ) with prior anti-PD-1 or anti-PD-L1 based treated tumour.
* Cohort 2 Patients with secondary resistance to anti-PD-1 or anti-PD-L1 based therapy: Any advanced or metastatic solid tumour with previously anti-PD-1 or anti-PD-L1 based treatment who progressed after achieving benefit
* Cohort 3 Patients with primary resistance to anti-PD-1 or anti-PD-L1 based therapy: Select advanced or metastatic solid tumour types with previous anti-PD- 1/PD-L1 based treated tumour without achieving benefit.
* All patients must have measurable lesions according to RECIST v1.1
* Patient must agree to pre- and on-treatment tumour biopsies. If archived tumour tissue is available from the last treatment failure, sections may be supplied instead of a pre-treatment biopsy.

Module C:

* Histologically confirmed diagnosis of one of the following cohorts:

  * Cohort 1: GEC: Locally advanced, unresectable or metastatic gastric adenocarcinoma or GEC.
  * Cohort 2: Patients with secondary resistance to anti-PD-1 or anti-PD-L1 based therapy: Any advanced or metastatic solid tumour (excluding NSCLC and melanoma) with previously anti-PD-1 or anti-PD-L1 based treatment which progressed after achieving benefit.
  * Cohort 3: Patients with primary resistance to anti-PD-1 or anti-PD-L1 based therapy: Select advanced or metastatic solid tumour types with previous anti-PD-1/PD-L1 based treated tumour without achieving benefit.
  * Cohort 4: Locally advanced, unresectable or metastatic second line or greater, microsatellite stable (MSS) colorectal cancer.
  * Cohort 5: Advanced Endometrial cancer: Endometrial carcinoma that is pMMR (Mismatch Repair-Proficient)/MSS and is advanced, recurrent, or persistent and has relapsed or is refractory to curative therapy.
* All patients must have at least one measurable lesion according to RECIST v1.1
* Further inclusion criteria apply

Exclusion Criteria

Master Protocol:

* Any investigational treatment anti-tumour treatment within 4 weeks or within 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment.
* More than one anti-PD-(L)1-based treatment regimen prior to entering study study, more specifically defined in the modules. Note: once in a trial Module, patients may crossover to different Module if all other eligibility criteria are met.
* Major surgery ('major' according to the Investigator's assessment) performed within 12 weeks prior to first trial treatment or planned within 12 months after screening, e.g., hip replacement.
* Known history of severe hypersensitivity reactions to other mAbs or known hypersensitivity to the trial drugs or their excipients.
* Presence of central nervous system (CNS) metastases, unless treated and asymptomatic and off corticosteroids and/or anticonvulsant therapy for at least 2 weeks prior to start of treatment.
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment.
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy. Patients who were permanently discontinued from previous anti-PD-1 or anti-PD-L1 therapy because of an immune-related adverse event (irAE).

Module A:

- Previous treatment with an anti-LAG-3 Agent

Module C:

* Unresolved, Grade >1 toxicity before the start of treatment with the study drug except for hair loss (alopecia) and hypothyroidism that requires thyroid hormone supplements but is asymptomatic under therapy.
* Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > New York Heart Association [NYHA] II)
* History of severe haemorrhagic or thromboembolic event in the past 12 months
* Known inherited predisposition to bleeding or to thrombosis, in the opinion of the investigator - Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - University of California San Diego, La Jolla, California
  - Florida Cancer Specialists-Fort Myers-52980, Fort Myers, Florida
  - Florida Cancer Specialists-Saint Petersburg-52979, St. Petersburg, Florida
  - Florida Cancer Specialists-Sarasota-61670, Tallahassee, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Indiana University, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Oklahoma University School of Community Medicine, Oklahoma City, Oklahoma
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC-Nashville-52568, Nashville, Tennessee
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College Hospital, London
  - Guy's Hospital, London
  - Sarah Cannon Research Institute, London, London

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases(in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Platform trial evaluating the safety and efficacy of different ezabenlimab (BI 754091) treatment regimens on patients with different types of advanced or metastatic tumors: module C evaluated the efficacy and safety of ezabenlimab (BI 754091) in combination with BI 836880 and module A evaluated the efficacy and safety of ezabenlimab (BI 754091) in combination with BI 754111.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Started (Treated with study drugs) | 28 | 30 | 28 | 30 | 18 | 2 | 33 | 42
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 28 | 30 | 28 | 30 | 18 | 2 | 33 | 42
Not completed — Other than listed | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 1 | 2 | 4 | 0 | 1 | 0 | 1 | 0
Not completed — Consent withdrawal | 1 | 2 | 0 | 4 | 4 | 0 | 1 | 1
Not completed — Adverse Event | 4 | 4 | 2 | 4 | 4 | 1 | 5 | 3
Not completed — Progressive disease | 21 | 20 | 22 | 22 | 8 | 1 | 25 | 37

BASELINE CHARACTERISTICS:
Population: Treated set: all patients treated with at least one dose of trial medications.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients | Total
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18 | 2 | 33 | 42 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (10.7) | 63.2 (13.3) | 60.6 (10.9) | 57.7 (13.5) | 67.8 (11.3) | 61.0 (14.1) | 68.6 (7.2) | 64.9 (10.4) | 66.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 7 | 13 | 18 | 1 | 14 | 22 | 93
  Male | 20 | 20 | 21 | 17 | 0 | 1 | 19 | 20 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 4 | 10
  Not Hispanic or Latino | 8 | 16 | 22 | 27 | 17 | 2 | 33 | 37 | 162
  Unknown or Not Reported | 20 | 12 | 5 | 0 | 1 | 0 | 0 | 1 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 10
  Black or African American | 0 | 0 | 1 | 1 | 2 | 0 | 4 | 2 | 10
  Other | 20 | 12 | 5 | 1 | 1 | 0 | 0 | 3 | 42
  White | 7 | 16 | 20 | 25 | 13 | 2 | 28 | 36 | 147

OUTCOME MEASURES:

1. Secondary Outcome: [Module C] Duration of Response (DoR)
Description: Duration of response (DoR) was defined as the time from first documented complete response (CR) or partial response (PR) (RECIST v1.1) among patients with objective response (OR), according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1). Complete response (CR) was defined as the disappearance of all target lesions and partial response (PR) was defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. DoR parameters were calculated based on Kaplan-Meier estimation. The analysis was performed on the unconfirmed OR.
Time Frame: From first documented CR or PR (RECIST v1.1) until the earlier of disease progression or death. Up to 174.6 weeks.
Population: Treated set of the module C: all patients treated with at least one dose of trial medications. Only patients that had an unconfirmed OR were included in the analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 4 | 9 | 2 | 2 | 8
Weeks | 105.95 [12.3 to 174.6] | 30.90 [6.4 to 81.3] | 8.50 [8.4 to 8.6] | 25.00 [12.1 to 37.9] | 47.30 [6.1 to 143.1]

2. Secondary Outcome: [Module C] Disease Control (DC)
Description: Disease Control (DC) defined as the percentage of patients with best overall response of complete response (CR), partial response (PR), or stable disease (SD), assessed by the investigator according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1). CR was defined as the disappearance of all target lesions, PR was defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study, and PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From first drug administration until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy. Up to approximately 188.3 weeks.
Population: Treated set of module C: all patients treated with at least one dose of trial medications.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18
percentage of participants | 57.1 [37.2 to 75.5] | 73.3 [54.1 to 87.7] | 42.9 [24.5 to 62.8] | 56.7 [37.4 to 74.5] | 77.8 [52.4 to 93.6]

3. Secondary Outcome: [Module C] Disease Control (DC) - Bayesian Hierarchical Model
Description: Disease Control (DC), defined as the disease control rate (DCR) of participants with best overall response of complete response (CR), partial response (PR), or stable disease (SD), assessed by the investigator according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1). CR was defined as the disappearance of all target lesions, PR was defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study, and PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The estimated DCR is presented by the posterior medians of the bayesian hierarchical model and by the correspondent credible intervals.
Time Frame: as for outcome 2
Population: Treated set of module C: all patients treated with at least one dose of trial medications.
Measure: Median (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18
percentage of participants | NA [NA to NA] — Posterior median = 64.7 97.5% credible interval = (45.4, 77.8) | NA [NA to NA] — Posterior median = 70.4 97.5% credible interval = (56.7, 83.8) | NA [NA to NA] — Posterior median = 44.7 97.5% credible interval = (29.1, 59.8) | NA [NA to NA] — Posterior median = 57.5 97.5% credible interval = (42.1, 71.5) | NA [NA to NA] — Posterior median = 82.2 97.5% credible interval = (66.7, 96.1)

4. Secondary Outcome: [Module C] Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from first treatment administration until progressive disease (PD), according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1), or death from any cause, whichever occurred earlier. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. PFS parameters were calculated based on Kaplan-Meier estimation.
Time Frame: From first drug administration until PD or death, whichever occurred earlier. Up to approximately 186.1 weeks.
Population: Treated set of module C: all patients treated with at least one dose of trial medications.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18
Weeks | 13.4 [6.1 to 33.7] | 29.1 [13.0 to 48.7] | 6.1 [5.7 to 12.1] | 12.6 [6.1 to 23.6] | 75.0 [24.9 to NA] — NA = not calculable due to insufficient number of participants with the event.

5. Secondary Outcome: [Module A] Duration of Response (DoR)
Description: as for outcome 1
Time Frame: From first documented CR or PR (RECIST v1.1) until the earlier of disease progression or death. Up to 63.6 weeks.
Population: Treated set of the module A: all patients treated with at least one dose of trial medications. Only patients that had an unconfirmed OR were included in the analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 0 | 3 | 8
Weeks |  | 12.30 [5.7 to 31.4] | 28.30 [0.1 to 63.6]

6. Secondary Outcome: [Module A] Disease Control (DC)
Description: as for outcome 2
Time Frame: From first drug administration until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy. Up to approximately 152.4 weeks.
Population: Treated set on module A: all patients treated with at least one dose of trial medications.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 2 | 33 | 42
percentage of participants | 0 [0.0 to 84.2] | 42.4 [25.5 to 60.8] | 45.2 [29.8 to 61.3]

7. Secondary Outcome: [Module A] Disease Control (DC) - Bayesian Hierarchical Model
Description: as for outcome 3
Time Frame: as for outcome 6
Population: Treated set on module A: all patients treated with at least one dose of trial medications.
Measure: Median (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 2 | 33 | 42
percentage of participants | NA [NA to NA] — Posterior median = 10.83 97.5 % credible interval = (1.7, 28.79) | NA [NA to NA] — Posterior median = 42.83 97.5 % credible interval = (28.86, 57.14) | NA [NA to NA] — Posterior median = 44.18 97.5 % credible interval = (31.57, 57.68)

8. Secondary Outcome: [Module A] Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from first treatment administration until progressive disease (PD), according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1), or death from any cause, whichever occurred earlier. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. PFS parameters were calculated based on Kaplan-Meier estimation. Progression free survival was collected, according to the clinical trial protocol until July 2021.
Time Frame: From first drug administration until PD, death, or cut-off date of July 2021, whichever occurred earlier. Up to approximately 104.7 weeks.
Population: Treated set of module A: all patients treated with at least one dose of trial medications.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 2 | 33 | 42
Weeks | 5.9 [5.7 to NA] — NA = not evaluable due to insufficient number of participants with event | 6.7 [5.9 to 11.9] | 8.9 [5.7 to 16.9]

9. Primary Outcome: [Module C] Objective Response (OR)
Description: Confirmed objective response (OR), defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), assessed by the investigator according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1). Complete response (CR) was defined as the disappearance of all target lesions and partial response (PR) was defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference.
Time Frame: as for outcome 2
Population: Treated set of the module C: all patients treated with at least one dose of trial medications.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18
percentage of participants | 14.3 [4.0 to 32.7] | 23.3 [9.9 to 42.3] | 0.0 [0.0 to 12.3] | 3.3 [0.1 to 17.2] | 44.4 [21.5 to 69.2]

10. Primary Outcome: [Module C] Objective Response (OR) - Bayesian Hierarchical Model
Description: Confirmed objective response (OR), defined as the objective response rate (ORR) of participants with best overall response of complete response (CR) or partial response (PR), assessed by the investigator according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1). Complete response (CR) was defined as the disappearance of all target lesions and partial response (PR) was defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. The estimated objective response rate is presented by the posterior medians of the Bayesian hierarchical model and by the correspondent credible intervals.
Time Frame: as for outcome 2
Population: Treated set of the module C: all patients treated with at least one dose of trial medications.
Measure: Median (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients
Number analyzed (Participants) | 28 | 30 | 28 | 30 | 18
percentage of participants | NA [NA to NA] — Posterior median = 11.95 97.5 % credible interval = (3.72, 25.31) | NA [NA to NA] — Posterior median = 20.21 97.5 % credible interval = (9.61, 36.1) | NA [NA to NA] — Posterior median = 2.75 97.5 % credible interval = (0.17, 10.15) | NA [NA to NA] — Posterior median = 5.26 97.5 % credible interval = (0.83, 14.87) | NA [NA to NA] — Posterior median = 36.13 97.5 % credible interval = (17.15, 59.63)

11. Primary Outcome: [Module A] Objective Response (OR)
Description: as for outcome 9
Time Frame: as for outcome 6
Population: Treated set of the module A: all patients treated with at least one dose of trial medications.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 2 | 33 | 42
percentage of participants | 0.0 [0.0 to 84.2] | 6.1 [0.7 to 20.2] | 9.5 [2.7 to 22.6]

12. Primary Outcome: [Module A] Objective Response (OR) - Bayesian Hierarchical Model
Description: as for outcome 10
Time Frame: as for outcome 6
Population: Treated set of the module A: all patients treated with at least one dose of trial medications.
Measure: Median (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
Number analyzed (Participants) | 2 | 33 | 42
percentage of participants | NA [NA to NA] — Posterior median = 9.69 97.5 % credible interval = (0.88, 35.04) | NA [NA to NA] — Posterior median = 8.23 97.5 % credible interval = (2.12, 18.91) | NA [NA to NA] — Posterior median = 6.67 97.5 % credible interval = (2.3, 16.02)

ADVERSE EVENTS:
Time Frame: Adverse event reporting and all-cause mortality: From first until last drug administration plus residual effect period (30 days). Up to approximately 192.6 weeks for module C and approximately 156.7 weeks for module A.
Description: Treated set: all patients treated with at least one dose of trial medications.
Groups:
- Module C, Cohort 3: 1ary Resistance Patients: Patients with select advanced or metastatic solid tumors with prior anti-PD-1- or anti-PD-L1-based treatment without achieving benefit ( stable disease duration of less than 4 months or progressive disease in less than 4 months while on treatment), were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
- Module C, Cohort 4: CRC Patients: Patients with locally advanced, unresectable or metastatic second-line or greater, microsatellite-stable colorectal cancer (CRC) without prior anti-PD-1- or anti-PD-L1-based treatment, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
- Module C, Cohort 5: EC Patients: Patients with advanced endometrial carcinoma (EC), excluding microsatellite instability-high or mismatch repair deficient types, who progressed following one line of chemotherapy, were not eligible for curative surgery or radiation, and had not been previously treated with anti-PD-1- or anti-PD-L1-based therapies, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 720 mg of BI 836880, intravenously, on Day 1 of 21-day cycles.
- Module A, Cohort 2: 2ary Resistance Patients: Patients with any advanced or metastatic solid tumors who had been previously treated with anti-PD-1 or anti-PD-L1-based therapies, and who progressed after achieving benefit (at least stable disease with a minimum duration of benefit of 6 months) and minimum treatment duration of 2 months without experiencing disease progression, were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
- Module A, Cohort 3: 1ary Resistance Patients: Patients with select advanced or metastatic solid tumor types, who have been previously treated with previous anti-PD-1 or anti-PD-L1-based therapies without achieving benefit (stable disease for less than 6 months or progressive disease in less than 6 months), were administered 240 mg of ezabenlimab (BI 754091), intravenously, on Day 1 of 21-day cycles, along 600 mg of BI 754111, intravenously, on Day 1 of 21-day cycles.
Arm/Group | Module C, Cohort 1: GEC Patients | Module C, Cohort 2: 2ary Resistance Patients | Module C, Cohort 3: 1ary Resistance Patients | Module C, Cohort 4: CRC Patients | Module C, Cohort 5: EC Patients | Module A, Cohort 1: GEC Patients | Module A, Cohort 2: 2ary Resistance Patients | Module A, Cohort 3: 1ary Resistance Patients
All-Cause Mortality (participants affected / at risk) | 24/28 | 20/30 | 22/28 | 17/30 | 4/18 | 0/2 | 29/33 | 32/42
Serious Adverse Events (participants affected / at risk) | 11/28 | 18/30 | 12/28 | 13/30 | 11/18 | 1/2 | 13/33 | 12/42
Other Adverse Events (participants affected / at risk) | 27/28 | 27/30 | 26/28 | 29/30 | 18/18 | 2/2 | 33/33 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Module C, Cohort 1: GEC Patients (N=28) | Module C, Cohort 2: 2ary Resistance Patients (N=30) | Module C, Cohort 3: 1ary Resistance Patients (N=28) | Module C, Cohort 4: CRC Patients (N=30) | Module C, Cohort 5: EC Patients (N=18) | Module A, Cohort 1: GEC Patients (N=2) | Module A, Cohort 2: 2ary Resistance Patients (N=33) | Module A, Cohort 3: 1ary Resistance Patients (N=42)
ANAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BANDAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
IMMUNE THROMBOCYTOPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE LEFT VENTRICULAR FAILURE (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (CARDIAC DISORDERS) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (CARDIAC DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CARDIAC ARREST (CARDIAC DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDITIS (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ADRENAL INSUFFICIENCY (ENDOCRINE DISORDERS) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
ASCITES (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
COLITIS (GASTROINTESTINAL DISORDERS) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
DIARRHOEA (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (GASTROINTESTINAL DISORDERS) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
ILEUS (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
IMMUNE-MEDIATED ENTEROCOLITIS (GASTROINTESTINAL DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LARGE INTESTINE PERFORATION (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NAUSEA (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
OESOPHAGEAL OBSTRUCTION (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OESOPHAGEAL PERFORATION (GASTROINTESTINAL DISORDERS) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PANCREATITIS (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RECTAL HAEMORRHAGE (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (GASTROINTESTINAL DISORDERS) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
DEATH (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DEVICE RELATED THROMBOSIS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FACE OEDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
IMPLANT SITE PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LOCALISED OEDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MALAISE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OEDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PYREXIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BILE DUCT STENOSIS (HEPATOBILIARY DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BILE DUCT STONE (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BILIARY OBSTRUCTION (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DRUG-INDUCED LIVER INJURY (HEPATOBILIARY DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC FAILURE (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERTRANSAMINASAEMIA (HEPATOBILIARY DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
JAUNDICE CHOLESTATIC (HEPATOBILIARY DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIVER INJURY (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ENCEPHALITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROINTESTINAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFECTED FISTULA (INFECTIONS AND INFESTATIONS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MENINGITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PHARYNGITIS BACTERIAL (INFECTIONS AND INFESTATIONS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (INFECTIONS AND INFESTATIONS) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
PNEUMONIA ASPIRATION (INFECTIONS AND INFESTATIONS) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
SEPSIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
VASCULAR DEVICE INFECTION (INFECTIONS AND INFESTATIONS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FALL (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
FEMUR FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HIP FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HUMERUS FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROCEDURAL PNEUMOTHORAX (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (INVESTIGATIONS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TROPONIN I INCREASED (INVESTIGATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERCALCAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOKALAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPONATRAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LACTIC ACIDOSIS (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYELODYSPLASTIC SYNDROME (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
TUMOUR ASSOCIATED FEVER (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TUMOUR THROMBOSIS (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
ENCEPHALOPATHY (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
SOMNOLENCE (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DELIRIUM (PSYCHIATRIC DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (RENAL AND URINARY DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
HAEMATURIA (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYDRONEPHROSIS (RENAL AND URINARY DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
IMMUNE-MEDIATED NEPHRITIS (RENAL AND URINARY DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NEPHRITIS (RENAL AND URINARY DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
URINARY RETENTION (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY TRACT OBSTRUCTION (RENAL AND URINARY DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PROSTATITIS (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ACUTE RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ASPIRATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DYSPNOEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
ORGANISING PNEUMONIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1
PNEUMOTHORAX (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
PULMONARY EMBOLISM (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DERMATITIS BULLOUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (VASCULAR DISORDERS) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 3
HAEMORRHAGE (VASCULAR DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (VASCULAR DISORDERS) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Module C, Cohort 1: GEC Patients (N=28) | Module C, Cohort 2: 2ary Resistance Patients (N=30) | Module C, Cohort 3: 1ary Resistance Patients (N=28) | Module C, Cohort 4: CRC Patients (N=30) | Module C, Cohort 5: EC Patients (N=18) | Module A, Cohort 1: GEC Patients (N=2) | Module A, Cohort 2: 2ary Resistance Patients (N=33) | Module A, Cohort 3: 1ary Resistance Patients (N=42)
ANAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 4 | 2 | 1 | 1 | 1 | 0 | 5 | 6
THROMBOCYTOPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
ATRIAL FIBRILLATION (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ATRIAL TACHYCARDIA (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TACHYCARDIA (CARDIAC DISORDERS) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
EAR DISCOMFORT (EAR AND LABYRINTH DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EAR PAIN (EAR AND LABYRINTH DISORDERS) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
HYPOACUSIS (EAR AND LABYRINTH DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERTHYROIDISM (ENDOCRINE DISORDERS) | 2 | 0 | 0 | 1 | 2 | 0 | 3 | 0
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 1 | 4 | 3 | 6 | 5 | 0 | 2 | 7
CONJUNCTIVOCHALASIS (EYE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PERIORBITAL OEDEMA (EYE DISORDERS) | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0
VISION BLURRED (EYE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
ABDOMINAL DISTENSION (GASTROINTESTINAL DISORDERS) | 1 | 3 | 0 | 3 | 2 | 0 | 2 | 0
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 8 | 2 | 2 | 4 | 3 | 0 | 3 | 4
ABDOMINAL PAIN UPPER (GASTROINTESTINAL DISORDERS) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1
ASCITES (GASTROINTESTINAL DISORDERS) | 2 | 2 | 1 | 2 | 0 | 0 | 1 | 1
COLITIS (GASTROINTESTINAL DISORDERS) | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 2 | 3 | 2 | 3 | 4 | 0 | 6 | 10
DIARRHOEA (GASTROINTESTINAL DISORDERS) | 9 | 6 | 5 | 5 | 8 | 1 | 7 | 4
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 2
DYSPHAGIA (GASTROINTESTINAL DISORDERS) | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 3
EPIGASTRIC DISCOMFORT (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FLATULENCE (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (GASTROINTESTINAL DISORDERS) | 0 | 0 | 1 | 3 | 2 | 0 | 2 | 0
GINGIVAL BLEEDING (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
GINGIVAL PAIN (GASTROINTESTINAL DISORDERS) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NAUSEA (GASTROINTESTINAL DISORDERS) | 5 | 7 | 3 | 11 | 7 | 2 | 12 | 9
ORAL DISCOMFORT (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
PANCREATITIS ACUTE (GASTROINTESTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
STOMATITIS (GASTROINTESTINAL DISORDERS) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2
TOOTHACHE (GASTROINTESTINAL DISORDERS) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
VOMITING (GASTROINTESTINAL DISORDERS) | 4 | 6 | 2 | 10 | 7 | 1 | 5 | 5
ADMINISTRATION SITE REACTION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2
EARLY SATIETY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FACE OEDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 7 | 8 | 8 | 11 | 8 | 1 | 12 | 19
INFLUENZA LIKE ILLNESS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2
OEDEMA PERIPHERAL (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 | 6 | 4 | 12 | 6 | 0 | 3 | 4
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2
PYREXIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 2 | 1 | 1 | 3 | 0 | 4 | 5
SENSATION OF FOREIGN BODY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLECYSTITIS (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERTRANSAMINASAEMIA (HEPATOBILIARY DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (INFECTIONS AND INFESTATIONS) | 3 | 1 | 1 | 2 | 4 | 0 | 0 | 0
CYSTITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FOLLICULITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FUNGAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
GASTROINTESTINAL VIRAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
GROIN ABSCESS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
INFLUENZA (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
ORAL HERPES (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA (INFECTIONS AND INFESTATIONS) | 1 | 0 | 2 | 1 | 2 | 0 | 4 | 1
RHINITIS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SINUSITIS (INFECTIONS AND INFESTATIONS) | 1 | 0 | 3 | 1 | 1 | 0 | 3 | 0
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
TOOTH ABSCESS (INFECTIONS AND INFESTATIONS) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 5
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 3 | 3 | 3 | 4 | 5 | 0 | 6 | 5
CORNEAL ABRASION (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FALL (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 3 | 1 | 3 | 0 | 0 | 1 | 3
INFUSION RELATED REACTION (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 4 | 1 | 1 | 3 | 2 | 0 | 3 | 1
MUSCLE STRAIN (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SPINAL COMPRESSION FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
WOUND (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 1 | 1 | 2 | 2 | 3 | 0 | 2 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 1 | 0 | 2 | 4 | 1 | 0 | 1 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1
BLOOD BILIRUBIN INCREASED (INVESTIGATIONS) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
BLOOD CREATININE INCREASED (INVESTIGATIONS) | 1 | 4 | 3 | 6 | 1 | 0 | 2 | 2
BLOOD UREA INCREASED (INVESTIGATIONS) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
PLATELET COUNT DECREASED (INVESTIGATIONS) | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 0
RED BLOOD CELL COUNT INCREASED (INVESTIGATIONS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VITAMIN D DECREASED (INVESTIGATIONS) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
WEIGHT DECREASED (INVESTIGATIONS) | 5 | 2 | 4 | 13 | 3 | 0 | 7 | 7
WEIGHT INCREASED (INVESTIGATIONS) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1
DECREASED APPETITE (METABOLISM AND NUTRITION DISORDERS) | 3 | 5 | 1 | 5 | 5 | 0 | 8 | 9
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 1 | 2 | 2 | 2 | 3 | 1 | 7 | 5
HYPERCALCAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
HYPERKALAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 1
HYPERLIPIDAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
HYPERURICAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 1
HYPOALBUMINAEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 1
HYPOCALCAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 0
HYPOKALAEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 | 2 | 2 | 5 | 0 | 1 | 0 | 0
HYPOMAGNESAEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 0
HYPONATRAEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0
VITAMIN B12 DEFICIENCY (METABOLISM AND NUTRITION DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5 | 5 | 5 | 2 | 2 | 0 | 8 | 5
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5 | 1 | 1 | 0 | 2 | 0 | 3 | 6
FLANK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 1 | 0 | 1 | 2 | 0 | 4 | 0
GROIN PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
MUSCLE SPASMS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 2 | 0 | 2 | 1 | 0 | 4 | 2
MUSCULAR WEAKNESS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 2
MUSCULOSKELETAL CHEST PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 3
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 2 | 4 | 0 | 1 | 0 | 1 | 0
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 0 | 1 | 1 | 4 | 0 | 4 | 3
PAIN IN JAW (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
APHASIA (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (NERVOUS SYSTEM DISORDERS) | 1 | 2 | 0 | 1 | 3 | 0 | 6 | 4
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1
HEADACHE (NERVOUS SYSTEM DISORDERS) | 2 | 4 | 2 | 2 | 4 | 0 | 6 | 3
MEMORY IMPAIRMENT (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
NEUROPATHY PERIPHERAL (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PARALYSIS RECURRENT LARYNGEAL NERVE (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
DEVICE DISLOCATION (PRODUCT ISSUES) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANXIETY (PSYCHIATRIC DISORDERS) | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 1
CONFUSIONAL STATE (PSYCHIATRIC DISORDERS) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3
DEPRESSION (PSYCHIATRIC DISORDERS) | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1
INSOMNIA (PSYCHIATRIC DISORDERS) | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1
DYSURIA (RENAL AND URINARY DISORDERS) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
HAEMATURIA (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 1
NEPHROLITHIASIS (RENAL AND URINARY DISORDERS) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
NOCTURIA (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
POLLAKIURIA (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
PROTEINURIA (RENAL AND URINARY DISORDERS) | 1 | 1 | 0 | 5 | 1 | 0 | 0 | 0
URINARY INCONTINENCE (RENAL AND URINARY DISORDERS) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 3 | 0 | 6 | 5 | 1 | 4 | 10
DYSPHONIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 1
DYSPNOEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 | 2 | 5 | 2 | 0 | 0 | 6 | 4
DYSPNOEA EXERTIONAL (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2
HAEMOTHORAX (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LARYNGEAL PAIN (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NASAL CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1
OROPHARYNGEAL PAIN (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 2
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 2
RHINITIS ALLERGIC (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
RHINORRHOEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
SINUS CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
HAND DERMATITIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 | 1 | 2 | 5 | 2 | 0 | 1 | 3
RASH (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 1
RASH ERYTHEMATOUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 3
RASH PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RASH PRURITIC (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HOT FLUSH (VASCULAR DISORDERS) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
HYPERTENSION (VASCULAR DISORDERS) | 3 | 9 | 6 | 8 | 7 | 0 | 1 | 1
HYPOTENSION (VASCULAR DISORDERS) | 0 | 0 | 3 | 0 | 0 | 0 | 6 | 0
LYMPHOEDEMA (VASCULAR DISORDERS) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (6):
  • Study Protocol: Study Protocol - Master (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/Prot_002.pdf
  • Study Protocol: Study Protocol - Module C (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/Prot_001.pdf
  • Study Protocol: Study Protocol - Module A (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/Prot_000.pdf
  • Statistical Analysis Plan: Statistical analysis Plan - Module A (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/SAP_004.pdf
  • Statistical Analysis Plan: Statistical analysis Plan - Module C (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/SAP_005.pdf
  • Statistical Analysis Plan: Statistical analysis Plan - Master (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03697304/SAP_003.pdf